CLINICAL TRIAL: NCT03195608
Title: Using Advanced Driver Assistance Systems (ADAS) as an Intervention Strategy for Drivers With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Liliana Alvarez Jaramillo, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 109272
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Driving Impaired
Keywords: In-vehicle technologies; Parkinson's disease; Driving performance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be masked regarding the pre or post-test status of the assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will complete a standardized battery of paper and pencil and computer tests. Following these tests, participants will complete a baseline simulator driving assessment without any form of assistive technology. We will employ a CDS-200 driving simulator (DriveSafety Inc., Salt Lake City, UT). A trained blinded evaluator will observe the recorded drive and score the drive. After the baseline assessment, participants will engage in 3 intervention sessions (lasting 30 minutes each). During these sessions, the lane change assistance system will be introduced and participants will be taught how to use it. After the 3 sessions, participants will participate in a post-test, similar to the baseline assessment but with a different route within the simulated world. They will drive this new route with the assistive technology. One to two weeks after the post-test, participants will be invited to participate in a follow-up assessment (battery of tests and simulator assessment).
  Interventions: Device: Lane change assistance system
- Control (Active Comparator): Participants will complete a standardized battery of paper and pencil and computer tests. Following these tests, participants will complete a baseline simulator driving assessment without any form of assistive technology. We will employ a CDS-200 driving simulator (DriveSafety Inc., Salt Lake City, UT). A trained blinded evaluator will observe the recorded drive and score the drive. After the baseline assessment, participants will engage in 3 intervention sessions (lasting 30 minutes each). During these sessions, participants will drive the scenario and receive feedback from a trained evaluator regarding their live performance. No lane change assistance system will be utilized. After the 3 sessions, participants will participate in a post-test, similar to the baseline assessment but with a different route within the simulated world.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Device: Lane change assistance system — This study will investigate the feasibility and preliminary efficacy of a 6-session lane change ADAS-intervention on the simulated driving performance of individuals with mild to moderate PD. We anticipate that the use of lane change assist technology will decrease the number of driving errors in individuals with PD. As this is a feasibility study, we will evaluate: -recruitment capability and sample characteristics - data collection methods, procedures, and outcome measures - acceptability and suitability of the lane change assist technology intervention - preliminary efficacy The outcomes of this study will inform the design of a larger study, should such large-scale study be warranted.
  Arms: Intervention
Behavioral: Active Control — Participants will practice their driving on a driving simulator with feedback form a trained interventionist.
  Other Names: Simulator practice
  Arms: Control

SUMMARY:
Parkinson's disease (PD) impacts an individual's fitness to drive in a number of ways that increase the crash risk in this population. Current vehicle automation technologies are available, that although designed for the general public, may help drivers with PD stay on the roads longer and safer than currently possible. Using a driving simulator (a safe and cost-effective alternative with no impact on licensing for participants), this study will investigate the feasibility and preliminary efficacy of utilizing in-vehicle technology (i.e., a simulated lane change assistance system) to address critical driving errors in individuals with mild to moderate Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 21 years of age or older (as a feasibility study, this study will provide the opportunity to participate to those diagnosed with early onset PD)
* Have been diagnosed with Parkinson's disease by a neurologist or movement disorder specialist
* Currently hold a valid G driver's license
* Meet provincial visual acuity (20/50 binocular) and visual field (120 continuous along the horizontal meridian with both eyes examined together) requirements for driving
* Be proficient in English reading and speaking (self-reported).

Exclusion Criteria:

* Have any other neurological or psychiatric conditions that would interfere with full participation in the study
* Be taking psychotropic medication(s) that affect their mental and/or physical functioning

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in number of lane maintenance errors from baseline to post-test 1(4 weeks) and post-test 2 (6 weeks) | Baseline, 4 weeks, and 6 weeks
  Refers to the lateral position of the vehicle in the lane.
Change in number of visual scanning errors from baseline to post-test 1(4 weeks) and post-test 2 (6 weeks) | Baseline, 4 weeks, and 6 weeks
  Visual scanning is defined as eye movement and turning of the neck and head (e.g. glances, look sideways at an intersection, look at mirrors) to detect oncoming objects
Change in number of signalling errors from baseline to post-test 1(4 weeks) and post-test 2 (6 weeks) | Baseline, 4 weeks, and 6 weeks
  Refers to the proper use of turning signals during lane changes

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Alvarez, PhD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No